CLINICAL TRIAL: NCT01611844
Title: Optimization of Tuberculosis Intradermal Skin Test: TB Dermatest WP 3.1
Brief Title: Optimization of Tuberculosis Intradermal Skin Test
Acronym: TB Dermatest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2009.591
Record Dates: First submitted 2011-12-22; First posted 2012-06-05 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2013-07

CONDITIONS: Healthy Volunteers
Keywords: delayed-type hypersensitivity reaction to tuberculin intradermal injection; tuberculosis skin test; BD micro-needle; medical device; spectroscopy
MeSH Terms: interventions — Tuberculin Test

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical device : micro-needle BD 1.5 mm 30G (Experimental)
  Interventions: Device: Medical device : micro-needle BD 1.5 mm 30G drug:Tubertest® : tuberculin (purified protein derivative)
- Manthoux method: lance 26G X 16mm (Active Comparator)
  Interventions: Device: medical device: lance 26G X 16mm drug: Tubertest® : tuberculin (purified protein derivative)

INTERVENTIONS:
Device: Medical device : micro-needle BD 1.5 mm 30G drug:Tubertest® : tuberculin (purified protein derivative) — 2 intradermal injections are performed on each arm/bottom of the subject:
  * 1 intradermal injection of Tuberculin (5UI)
  * 1 intradermal injection of saline solution using Manthoux method or BD micro-needle. the method of injection is randomized: left or right
  Arms: Medical device : micro-needle BD 1.5 mm 30G
Device: medical device: lance 26G X 16mm drug: Tubertest® : tuberculin (purified protein derivative) — 2 intradermal injections are performed on each arm/bottom of the subject:
  * 1 intradermal injection of Tuberculin (5UI)
  * 1 intradermal injection of saline solution using Manthoux method or BD micro-needle. the method of injection is randomized: left or right
  Arms: Manthoux method: lance 26G X 16mm

SUMMARY:
The only test available for in vivo diagnosis of tuberculosis is the intradermal injection of tuberculin according to the Mantoux method (also named tuberculosis skin test or PPD skin test).

The tuberculin skin test is based on a delayed-type hypersensitivity skin reaction However, this test needs to be performed by trained personnel, presents problem of reproducibility, and its interpretation is not well standardized (measure in millimeters of skin induration 48 to 72 hours after the PPD skin test).

The new generation BD micro needle used in this study should solve the technical difficulties; intradermal administration of tuberculin could then be made by any personnel.

A non-invasive and objective instrumental method of reading the test will be also tested .

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years or over
* Tuberculosis skin test (PPD)
* positive : 5mm =<PPD<15mm (24 subjects)
* negative: PPD < 5mm (6 subjects)
* Negative Quantiferon test.
* Legal capacity to consent
* Subject had given written consent before his participation
* Subject accepting to participate in the second phase of the study with skin biopsies (24 subjects with positive PPD)
* Females of childbearing potential using an effective method of contraception, for at least 1 month before the beginning of the study and until 1 month after the end of their participation

Exclusion Criteria:

* Known allergy to tuberculin
* History of severe skin reaction to tuberculin with vesicle, ulceration, necrosis
* History of active tuberculosis
* Latent tuberculosis (positive Quantiferon test)
* Contact with a person having or having had active tuberculosis in the previous 3 months
* Chronic disease non-stabilized under treatment
* Immunosuppressive therapy or corticosteroids within 1 month before PPD skin tests
* Non-steroid anti-inflammatory drugs within 1 week before PPD skin tests
* Application on study areas of topical drugs containing corticoids or immunosuppressants within 1 week before PPD skin test
* Dermatological disease on study area
* Known allergy to local anesthetics
* Wound healing disorders
* Subject in an exclusion period or participating or planning to participate in another biomedical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
hypersensitivity reaction to tuberculin measured in millimeters of skin induration by comparing two methods of intradermal injection (Mantoux and BD micro-needle). [Phase 1] | 72 h

SECONDARY OUTCOMES:
spectroscopy instrumentation(non-invasive and objective method)to measure the PPD reaction | 72 h
define changes in the cutaneous immune system at various times (7h, 24h and 48 h), induced by intradermal microinjection of tuberculin, by histological, immunohistochemical and molecular analysis | 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GOUJON, MD, Principal Investigator — Centre Hospitalier Lyon Sud -Hospices Civils de Lyon
Locations (1):
- Unité de Recherche Clinique en Immunologie Lyon Sud (URCI-LS) et Service d'Immunologie clinique et allergologie-Centre Hospitalier Lyon Sud -Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Background] Diffuse Reflectance Spectroscopy: A clinical study of tuberculin skin tests reading Anne Koenig, Sophie Grande, Karima Dahel, Anne Planat-Chrétien, Vincent Poher, Catherine Goujon, Jean- Marc Dinten. Biomedical Applications of Light Scattering VII, 85920S (21 February 2013)